CLINICAL TRIAL: NCT02162407
Title: A Randomised, Three-period Crossover Trial in Healthy Subjects Investigating the Relationship Between the Pharmacodynamic Steady State and the Pharmacokinetic Steady State in the Interstitial Fluid Following iv Infusion of Insulin Detemir and Human Insulin Using Microperfusion Technique
Brief Title: A Trial Investigating the Relationship Between Pharmacodynamic and Interstitial Concentration for Insulin Detemir and Human Insulin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN304-1196
Record Dates: First submitted 2014-05-22; First posted 2014-06-12 (Estimated); Last update posted 2014-06-12 (Estimated); Status verified 2014-06

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Insulin detemir 60 pmol/kg/min (Experimental): Subjects will be randomised to one of six treatment sequences (the 3 test drugs given at 3 different trial days 7-28 days apart in randomised order)
  Interventions: Drug: insulin detemir
- Insulin detemir 120 pmol/kg/min (Experimental): Subjects will be randomised to one of six treatment sequences (the 3 test drugs given at 3 different trial days 7-28 days apart in randomised order)
  Interventions: Drug: insulin detemir
- Human insulin 6 pmol/kg/min (Active Comparator): Subjects will be randomised to one of six treatment sequences (the 3 test drugs given at 3 different trial days 7-28 days apart in randomised order)
  Interventions: Drug: human soluble insulin

INTERVENTIONS:
Drug: insulin detemir — Given as intravenous infusion (i.v.) over a period of 8 hours during euglycaemic clamp
  Arms: Insulin detemir 120 pmol/kg/min; Insulin detemir 60 pmol/kg/min
Drug: human soluble insulin — Given as intravenous infusion (i.v.) over a period of 8 hours during euglycaemic clamp
  Arms: Human insulin 6 pmol/kg/min

SUMMARY:
This study is conducted in Europe. The aim of this study is to estimate the relationship between pharmacodynamic and interstitial pharmacokinetic steady state following intravenous (i.v.) administration of insulin detemir and human soluble insulin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males between 19 and 50 years inclusive
* The subject must give signed informed consent before any trial related activity. (Trial related activities are any procedures that would not have been performed during the normal management of the subject)
* Body Mass Index (BMI) below 27 kg/m^2
* Fasting blood glucose maximum 6 mmol/l

Exclusion Criteria:

* Participation in any other clinical trial involving other investigational products within the last 3 months

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 1999-10; Primary Completion 1999-12 (Actual); Study Completion 1999-12 (Actual)

PRIMARY OUTCOMES:
Steady state glucose infusion rate (GIR) / interstitial insulin steady state concentration | 8 hours

SECONDARY OUTCOMES:
Steady state glucose infusion rate (GIR) | 8 hours
Steady state insulin interstitial concentration | 8 hours
Ratio of steady state serum insulin concentration to interstitial insulin concentration | 8 hours
Insulin concentration profiles | 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Graz, Austria

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com